CLINICAL TRIAL: NCT03763292
Title: Effect of Preoperative Information to Parents Before Ear-nose-throat Pediatric Surgery on the Parents' Preparedness for Anesthesia
Brief Title: Effect of Preoperative Information to Parents Before Ear-nose-throat Pediatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Helse Nord-Trøndelag HF (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: REK2018/1830
Record Dates: First submitted 2018-11-30; First posted 2018-12-04 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Anxiety; Consumer Satisfaction
Keywords: Parents; Patient Education as Topic; Preoperative Care; Pamphlets
MeSH Terms: conditions — Anxiety Disorders; Consumer Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Information brochure (Experimental): Intervention: The parents are given a specific information brochure that describes the procedures that the child is going through during anesthesia when it has been decided that the child is going to have the surgery.
  Interventions: Behavioral: Specific information brochure
- Information as usual (No Intervention): Information as usual, i.e. oral information about the procedures to parents when they arrive at the hospital with the child that is going to have the surgery.

INTERVENTIONS:
Behavioral: Specific information brochure — A purpose-designed brochure about anesthesia and surgery in the ear in children is developed by the investigators. This brochure has photos and describes the procedures the child is going through.
  Arms: Information brochure

SUMMARY:
Children who will have surgery and need anesthesia, and their parents are often anxious and show signs of stress and discomfort. A main reason for concern and anxiety is fear of anesthesia and surgery, and lack of knowledge of what is going to happen. The purpose of the study is to see if a specific preoperative information brochure aimed at the parents will make the parents feel better prepared for the procedures.

ELIGIBILITY:
Inclusion Criteria:

* Parents with children undergoing ear-nose-throat surgery in the study period

Exclusion Criteria:

* Parents who do not speak nor read Norwegian.
* Parents who do not want to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2020-07-03 (Actual); Study Completion 2020-07-03 (Actual)

PRIMARY OUTCOMES:
Satisfaction with information | 10 minutes
  Self-reported satisfaction with provided information on a 5 point Likert scale where 1 is less satisfied and 5 is high satisfaction (range 1-5). In total four questions (sum score range 4-20)
Preparedness for the operating room setting | 10 minutes
  Self-reported to what degree parents feel prepared as to what will happen before/during induction of anaesthesia on a 5 point Likert scale where 1 is less prepared and 5 is very well prepared (range 1-5). In total two questions (sum score range 2-10)

SECONDARY OUTCOMES:
Perceived Stress Score (PSS-14) | 10 minutes
  Self-reported perceived stress measured by 14 questions on a 5-point Likert scale where 1 is Never and 5 is very often. Range for the total score is 1-70.

CONTACTS AND LOCATIONS:
Overall Officials: Siri Forsmo, phd prof, Study Director — Norwegian University for Science and Technology
Locations (1):
- Sykehus Levanger, Levanger, Norway

IPD SHARING:
Plan to Share IPD: Yes
Anonymous participant data plotted in a SPSS file can be shared on request.
Supporting Information: Study Protocol
Time Frame: September 2019 - August 2024 (5 years)
Access Criteria: Request to contact persons.